CLINICAL TRIAL: NCT04317989
Title: The STUN (STop UNhealthy) Alcohol Use Now! Project: Using Practice Facilitation to Disseminate and Implement Patient-Centered Outcomes Research (PCOR) Evidence on Screening and Management of Unhealthy Alcohol Use in Primary Care
Brief Title: STUN (STop UNhealthy) Alcohol Use Now! Implementing Evidence-Based Services for Unhealthy Alcohol Use in Primary Care
Acronym: STUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-1853; 1R18HS027078-01 (AHRQ)
Record Dates: First submitted 2020-03-16; First posted 2020-03-23 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2023-11

CONDITIONS: Risky Health Behavior; Drinking, Alcohol; Alcohol Use Disorder; Drinking, Binge; Drinking Excessive
Keywords: Alcohol, Screening, Counseling, Primary Care
MeSH Terms: conditions — Health Risk Behaviors; Alcohol Drinking; Alcoholism; Binge Drinking

STUDY DESIGN:
Intervention Model Description: This trial will evaluate the effect of primary care practice facilitation on evidence-based screening, counseling, and Medication-Assisted Treatment (MAT). Practices are considered the participants; the intervention is conducted on the practice level. All enrolled practices receive the practice facilitation intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Practice Facilitation (Experimental): All enrolled practices will receive practice facilitation for the duration of the intervention period.
  Interventions: Other: Practice Facilitation

INTERVENTIONS:
Other: Practice Facilitation — 1. Implementing evidence-based protocols and the use of clinical algorithms (for screening, counseling, referral, and MAT) to engage the entire clinical team in a high standard delivery of care.
  2. Promoting a strong use of decision support tools and templates to support the practice workflow.
  3. Optimizing the use of the electronic health record (EHR) to pull clinical data on a monthly basis to guide the change process.
  4. Developing patient registries (e.g., for those identified to have AUD) to identify needed care
  5. Proactive, team-based care with assigned roles and responsibilities to prepare the clinical team to develop needed care and engage patients throughout the entire visit process.
  6. Enhancing the understanding of available counseling and referral resources to ensure that practices are confident that they have appropriate evidence-based intervention options.

SUMMARY:
STUN Alcohol Use Now is an intervention designed to use primary care practice support services (practice facilitation) to help small to medium-size practices (10 or fewer providers) identify and provide services for people with unhealthy alcohol use. The original recruitment goal was 135 primary care practices in North Carolina, which we were unable to meet due to pandemic-related barriers.

DETAILED DESCRIPTION:
STUN Alcohol Use Now is an intervention designed to use primary care practice support services (practice facilitation or PF) to help small to medium-size practices (10 or fewer providers) identify and provide services for people with unhealthy alcohol use. 135 primary care practices in North Carolina will be recruited.

Specific Aim 1 will evaluate the effect of PF on uptake of evidence-based screening and brief intervention (SBI) for unhealthy alcohol use. The investigators hypothesize that PF will increase screening for unhealthy alcohol use and provision of brief counseling. The secondary hypothesis is that practice-level and contextual factors (capacity for quality improvement, organizational readiness to implement change, and implementation climate) will moderate the effect of PF on use of evidence-based screening and brief intervention (SBI) for unhealthy alcohol use.

Specific Aim 2 will evaluate whether PF increases provision, among those identified as having an alcohol use disorder (AUD), provision of medication assisted treatment (MAT) or referral to specialty care.

Aim 3 (effect of providing embedded telehealth services) will not be evaluated due to lower enrollment than anticipated and delayed data collection (both related to the COVID-19 pandemic) which have prevented randomization among practices with slower uptake of SBI after 6 months of PF.

In Aim 4 the investigators will evaluate the effect of PF on the implementation of clinical practice and office systems changes to improve evidence-based SBI and MAT. The primary hypothesis is that PF will increase implementation of clinical practice and office systems changes to improve evidence-based SBI and MAT. The secondary hypotheses are that (a) practice capacity for quality improvement (QI), organizational readiness to implement change, and contextual factors will moderate the effect of PF on the implementation of clinical practice and office systems changes and (b) embedded telehealth services will increase implementation of clinical practice and office systems changes among practices with slower uptake.

ELIGIBILITY:
Inclusion Criteria:

* Small-to-medium sized primary care practices (10 or fewer providers) in North Carolina

Exclusion Criteria:

* Practices with fewer than 100 adult patients (18+ years) or more than 10 providers;
* practices unwilling to implement evidence-based screening and management of patients with unhealthy alcohol use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Number of adults screened for unhealthy alcohol use | 18 months
  number aged 18 or older who were screened with a validated tool for unhealthy alcohol use
Number of adults screened for unhealthy alcohol use | 12 months
  number aged 18 or older who were screened with a validated tool for unhealthy alcohol use
Number of adults screened for unhealthy alcohol use | 6 months
  number aged 18 or older who were screened with a validated tool for unhealthy alcohol use
Percent of adults screened for unhealthy alcohol use | 18 months
  percent of those aged 18 or older who were screened with a validated tool for unhealthy alcohol use
Percent of adults screened for unhealthy alcohol use | 12 months
  percent of those aged 18 or older who were screened with a validated tool for unhealthy alcohol use
Percent of adults screened for unhealthy alcohol use | 6 months
  percent of those aged 18 or older who were screened with a validated tool for unhealthy alcohol use

SECONDARY OUTCOMES:
Number of adults with a positive screen for unhealthy alcohol use | 18 months
  Of those aged 18 or older who were screened for unhealthy alcohol use, number who had a positive initial screening result
Number of adults with a positive screen for unhealthy alcohol use | 12 months
  Of those aged 18 or older who were screened for unhealthy alcohol use, number who had a positive initial screening result
Number of adults with a positive screen for unhealthy alcohol use | 6 months
  Of those aged 18 or older who were screened for unhealthy alcohol use, number who had a positive initial screening result
Percent of adults with a positive screen for unhealthy alcohol use | 18 months
  Of those aged 18 or older who were screened for unhealthy alcohol use, percentage who had a positive initial screening result
Percent of adults with a positive screen for unhealthy alcohol use | 12 months
  Of those aged 18 or older who were screened for unhealthy alcohol use, percentage who had a positive initial screening result
Percent of adults with a positive screen for unhealthy alcohol use | 6 months
  Of those aged 18 or older who were screened for unhealthy alcohol use, percentage who had a positive initial screening result
Number of adults provided with brief counseling for risky drinking | 18 months
  Of those aged 18 or older who were identified as having unhealthy alcohol use, number who received brief counseling (based on documentation in the medical record)
Number of adults provided with brief counseling for risky drinking | 12 months
  Of those aged 18 or older who were identified as having unhealthy alcohol use, number who received brief counseling (based on documentation in the medical record)
Number of adults provided with brief counseling for risky drinking | 6 months
  Of those aged 18 or older who were identified as having unhealthy alcohol use, number who received brief counseling (based on documentation in the medical record)
Percent of adults provided with brief counseling for risky drinking | 18 months
  Of those aged 18 or older who were identified as having unhealthy alcohol use, percentage who received brief counseling (based on documentation in the medical record)
Percent of adults provided with brief counseling for risky drinking | 12 months
  Of those aged 18 or older who were identified as having unhealthy alcohol use, percentage who received brief counseling (based on documentation in the medical record)
Percent of adults provided with brief counseling for risky drinking | 6 months
  Of those aged 18 or older who were identified as having unhealthy alcohol use, percentage who received brief counseling (based on documentation in the medical record)
Number of adults identified as having alcohol use disorder (AUD) | 18 months
  After screening, number of adult patients identified to have AUD (based on documented ICD diagnoses of AUD)
Number of adults identified as having alcohol use disorder (AUD) | 12 months
  After screening, number of adult patients identified to have AUD (based on documented ICD diagnoses of AUD)
Number of adults identified as having alcohol use disorder (AUD) | 6 months
  After screening, number of adult patients identified to have AUD (based on documented ICD diagnoses of AUD)
Percent of adults identified as having alcohol use disorder (AUD) | 18 months
  After screening, percentage of adult patients screened who were identified to have AUD (based on documented ICD diagnoses of AUD)
Percent of adults identified as having alcohol use disorder (AUD) | 12 months
  After screening, percentage of adult patients screened who were identified to have AUD (based on documented ICD diagnoses of AUD)
Percent of adults identified as having alcohol use disorder (AUD) | 6 months
  After screening, percentage of adult patients screened who were identified to have AUD (based on documented ICD diagnoses of AUD)
Number of adults prescribed pharmacotherapy for AUD | 18 months
  After screening, number of adult patients with AUD who receive evidence-based pharmacotherapy with naltrexone, acamprosate, disulfiram, or topiramate
Number of adults prescribed pharmacotherapy for AUD | 12 months
  After screening, number of adult patients with AUD who receive evidence-based pharmacotherapy with naltrexone, acamprosate, disulfiram, or topiramate
Number of adults prescribed pharmacotherapy for AUD | 6 months
  After screening, number of adult patients with AUD who receive evidence-based pharmacotherapy with naltrexone, acamprosate, disulfiram, or topiramate
Percent of adults with AUD who were prescribed pharmacotherapy for AUD | 18 months
  After screening, percent of adult patients identified as having AUD who receive evidence-based pharmacotherapy with naltrexone, acamprosate, disulfiram, or topiramate
Percent of adults with AUD who were prescribed pharmacotherapy for AUD | 12 months
  After screening, percent of adult patients identified as having AUD who receive evidence-based pharmacotherapy with naltrexone, acamprosate, disulfiram, or topiramate
Percent of adults with AUD who were prescribed pharmacotherapy for AUD | 6 months
  After screening, percent of adult patients identified as having AUD who receive evidence-based pharmacotherapy with naltrexone, acamprosate, disulfiram, or topiramate
Number of adults with AUD referred to specialty care for AUD | 18 months
  After screening, number of adult patients identified as having AUD who are referred to specialty care (e.g., psychiatry, CBT, motivational enhancement therapy, 12-step programs)
Number of adults with AUD referred to specialty care for AUD | 12 months
  After screening, number of adult patients identified as having AUD who are referred to specialty care (e.g., psychiatry, CBT, motivational enhancement therapy, 12-step programs)
Number of adults with AUD referred to specialty care for AUD | 6 months
  After screening, number of adult patients identified as having AUD who are referred to specialty care (e.g., psychiatry, CBT, motivational enhancement therapy, 12-step programs)
Percent of adults with AUD referred to specialty care for AUD | 18 months
  After screening, percentage of adults identified as having AUD who are referred to specialty care (e.g., psychiatry, CBT, motivational enhancement therapy, 12-step programs)
Percent of adults with AUD referred to specialty care for AUD | 12 months
  After screening, percentage of adults identified as having AUD who are referred to specialty care (e.g., psychiatry, CBT, motivational enhancement therapy, 12-step programs)
Percent of adults with AUD referred to specialty care for AUD | 6 months
  After screening, percentage of adults identified as having AUD who are referred to specialty care (e.g., psychiatry, CBT, motivational enhancement therapy, 12-step programs)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Jonas, MD, MPH, Principal Investigator — Ohio State University; Darren Dewalt, MD, MPH, Principal Investigator — UNC Chapel Hill
Locations (7):
- United States (7):
  - Mountain AHEC, Asheville, North Carolina
  - Charlotte AHEC, Charlotte, North Carolina
  - Greensboro AHEC, Greensboro, North Carolina
  - Eastern AHEC, Greenville, North Carolina
  - Wake AHEC, Raleigh, North Carolina
  - Area L AHEC, Rocky Mount, North Carolina
  - Southeast AHEC, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jonas DE, Barclay C, Grammer D, Weathington C, Birken SA, DeWalt DA, Shoenbill KA, Boynton MH, Mackey M, Riley S, Cykert S. The STUN (STop UNhealthy) Alcohol Use Now trial: study protocol for an adaptive randomized trial on dissemination and implementation of screening and management of unhealthy alcohol use in primary care. Trials. 2021 Nov 16;22(1):810. doi: 10.1186/s13063-021-05641-7. PMID 34784953

DOCUMENTS (1):
  • Informed Consent Form (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT04317989/ICF_000.pdf